CLINICAL TRIAL: NCT05459077
Title: Addressing Barriers to Anti-hypertensive Medication Adherence Among Persons Living With HIV Who Have Achieved Viral Suppression
Brief Title: Addressing Barriers to Anti-hypertensive Medication Adherence Among PLWH Who Have Achieved Viral Suppression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00108808
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Hypertension; HIV-1-infection
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Aim 3B group will participate in an adapted intervention related to blood pressure management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aim 3B (Other): This aim will evaluate the feasibility and acceptability of the adapted health care delivery intervention to improve anti-hypertensive medication adherence and blood pressure control in persons living with HIV at 24 weeks.
  Interventions: Behavioral: Hypertension control through education and monitoring

INTERVENTIONS:
Behavioral: Hypertension control through education and monitoring — Enrollment of 60 PLWH ≥18 years old receiving care at the Duke ID clinic who have achieved HIV viral suppression who take antihypertensive medication and have uncontrolled blood pressure. Subjects will have be given educational materials, blood pressure monitors to use and report findings, follow up with study coordinator and communication with subject's HIV provider in order to maximize blood pressure control..

SUMMARY:
Among those with hypertension, persons living with HIV (PWH) have a 50% higher risk of incident myocardial infarction compared to the general population, and they often fail to meet evidence-based treatment goals for hypertension. An important contributing factor for insufficient blood pressure control is non-adherence to antihypertensive medications. Research on medication adherence for PWH has largely focused on antiretroviral therapy adherence with limited focus on adherence to other non-AIDS condition medications.

With a large proportion of PWH in the U.S. achieving viral suppression, providers may now have an opportunity to focus on the management of non-AIDS conditions like hypertension. However, because PWH who have achieved suppression have reduced clinic encounters (once or twice a year) there is potential loss of opportunity to effectively monitor and intensify hypertension treatment as needed an important opportunity to focus on preventing cardiovascular disease. CVD and other non-AIDS comorbidities.

The study's overarching goal is to improve the hypertension outcomes for PWH on suppressive ART to reduce cardiovascular disease risk. In this study, we will identify and evaluate healthcare and patient-level factors that must be addressed in an intervention to increase hypertension medication adherence for PWH who have achieved viral suppression. We will use these factors to tailor an intervention and assess the feasibility and acceptability at the Duke ID clinic.

DETAILED DESCRIPTION:
The study is divided into 5 separate groups, Aim 1A, Aim 1B, Aim 2, Aim 3A and Aim 3B. Aims 1A and 1B will identify and evaluate patient-level factors that must be addressed in an intervention to increase hypertension medication adherence for (persons living with HIV) PWH who have achieved viral suppression. Aim 2 will identify HIV providers' practice norms after their patients achieve viral suppression and explore barriers faced in monitoring and managing patient adherence to antihypertensive medications to inform an intervention aimed at increasing antihypertensive medication adherence. Aim 3A will adapt the health care delivery intervention components to the Duke ID clinic context with key stakeholder input and data from Aims 1 and 2. Aim 3B will evaluate the feasibility and acceptability of the adapted health care delivery intervention to improve anti-hypertensive medication adherence and BP control in PWH at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

Aims 1A and 1B

* Age ≥18 years
* Confirmed HIV+ diagnosis
* Undetectable HIV viral load: defined as the most recent HIV viral load <200 copies/mL checked within the past year (assessed via chart abstraction)
* Hypertension diagnosis in medical records
* Taking an antihypertensive medication
* Receiving care at the Duke HIV clinic

Aim 2

* HIV providers including infectious disease physicians, internists or advance practice practitioners who have a patient pool of PLWH under their care in the last 6 months.

Aim 3A

* Stakeholders composed of willing participants recruited from the Duke ID clinic and may include, HIV providers, clinic directors, nurses, pharmacists, social workers, people living with HIV who have hypertension and take antihypertensive medications, and representatives of the community advisory boards, and any other key stakeholders.

Aim 3 B

* Age ≥18 years
* Confirmed HIV+ diagnosis
* Receiving care at the Duke ID clinic
* Achievement of HIV suppression defined as having HIV-1 RNA <200 copies/ml
* Take antihypertensive medications
* Uncontrolled BP over a 12 months period defined by participants with systolic BP>130mmHg on ≥ 2 occasions in the past 12 months as indicated in the individual patient's electronic medical records

Exclusion Criteria:

Aims 1A, 1B and 3B

* Severely hearing or speech impaired, or other disability that would limit participation in the intervention components
* In a nursing home and/or receiving in-patient psychiatric care
* Terminal illness with life expectancy < 4 months
* No reliable access to a telephone
* Pregnant, breast-feeding, or planning a pregnancy during the study period
* Planning to move out of the area in the next 6 months
* Non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by enrollment | 1 year
  Number of participants enrolled divided by total number of eligible patients in Duke Clinic 1K
Acceptability of nurse managed adherence strategy | Week 24
  Intervention Measure (Likert scale 1 completely disagree to 5 completely agree)
Usefulness of contact with nurse | Week 24
  Intervention Measure (Likert scale 1 completely disagree to 5 completely agree)
Subject's evaluation regarding ease of use of blood pressure machine | Week 24
  Intervention Measure (Likert scale 1 completely disagree to 5 completely agree)
Subject's evaluation of ease of the completion of blood pressure logs | Week 24
  Intervention Measure (Likert scale 1 completely disagree to 5 completely agree)

SECONDARY OUTCOMES:
Total number of telephone contacts | Week 24
Duration of time to reduce elevated BP to an under-control reading | Week 24
Total number of specialty referrals | Week 24
Number of anti-hypertensive medication changes | Week 24
Change in subject's self report of anti-hypertensive medication adherence | Baseline and Week 24
  Adherence to Hypertension and Medication Scales (Likert scale strongly disagree to strongly agree and not at all to very much)
Change in systolic blood pressure measurements | Baseline and Week 24
  Comparison of baseline versus Week 24 visit measurements

CONTACTS AND LOCATIONS:
Overall Officials: Charles Muiruri, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No